CLINICAL TRIAL: NCT07065760
Title: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms
Brief Title: University of Utah PS-IDE: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cali Johnson (Other)
Responsible Party: Sponsor-Investigator, Cali Johnson, Assistant Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00185860
Record Dates: First submitted 2025-06-30; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Juxtarenal Abdominal Aortic Aneurysm
Keywords: physician modified endovascular graft; juxtarenal abdominal aortic aneurysm; PMEG; FEVAR; Endovascular Aortic Repair
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Intervention Model Description: Prospective, single center, nonrandomized, single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Physician Modified Endograft (Experimental): Surgical procedure to repair the juxtarenal abdominal aortic aneurysm, during which the physician-modified endovascular graft (PMEG) device will be used.
  Interventions: Device: Endovascular Aneurysm Repair with Physician Modified Endograft

INTERVENTIONS:
Device: Endovascular Aneurysm Repair with Physician Modified Endograft — The surgeon will make an incision to access the femoral artery and insert a thin wire to guide the catheter to the juxtarenal aortic aneurysm. The main graft will be modified by hand to match the participant's anatomy, then reloaded and guided through the artery to the aorta. Once in place, the graft will be deployed, and additional stents will be inserted into vital arteries that supply the kidneys and bowels. Two smaller grafts will be placed into the iliac arteries.This allows blood to flow to the target organs and legs, protecting the aneurysm from rupture. All catheters will then be removed, leaving the graft in place, and the incisions will be closed.

SUMMARY:
The purpose of this study is to assess the effects of a physician-modified endovascular graft (PMEG) for juxtarenal aortic aneurysms by collecting data on its performance. Participants in the study will undergo surgery to repair their juxtarenal aortic aneurysm using the PMEG device. After the surgery, participants will attend several follow-up visits to monitor their recovery and the device's effectiveness. These follow-up visits will take place at hospital discharge, then at 1 month, 6 months, 12 months, and once a year for up to 5 years after surgery.

DETAILED DESCRIPTION:
A juxtarenal aortic aneurysm is an aneurysm that occurs near the renal arteries, which bring blood to the kidneys. This research study will evaluate if the physician-modified endovascular graft (PMEG) is safe and effective in the treatment of juxtarenal aortic aneurysms. The PMEG device is an investigational device, which means it has not been approved by the FDA. The device is designed to create a pathway through the aneurysm for blood flow to the arteries, reducing the blood pressure that the aneurysm experiences. There are several types of endovascular devices depending on how big the aneurysm is, where the aneurysm is located in relation to the kidney, or other physical measurements of the blood vessels. The upper portion of the device, or stent graft, will include between one and four holes (fenestrations). The holes allow the device to be located above the renal arteries (the blood vessels that supply blood to the kidneys) without blocking the blood flow to them. Smaller grafts are then placed in the blood vessels to the kidneys, the intestines, and liver to be connected to the main aortic graft, allowing blood to flow to the organs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient has a juxtarenal abdominal aortic aneurysm that meets at least one of the following:

   1. An aneurysm with a maximum diameter of ≥ 5.5 cm for male (≥ 5.0 cm for female) or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
   2. Aneurysm with a history of growth > 0.5 cm in 6 months
   3. Saccular aneurysm deemed at significant risk for rupture
   4. Symptomatic aneurysm
   5. Ruptured aneurysm
5. Patient has patent iliac or femoral arteries, with or without the use of conduit, that will allow endovascular access with the physician modified endovascular graft.
6. Patient has a suitable non-aneurysmal proximal aortic neck of ≥ 2 mm inferior to the most distal renal artery ostium.
7. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥ 15mm. The resultant repair should preserve patency in at least one hypogastric artery.
8. Patient has a suitable non-aneurysmal proximal aortic neck diameter between 20 and 32 mm, averaged across the diameters at the Celiac, SMA, at the lowest patent renal artery and at the midpoint of the renal arteries.
9. Patient has suitable non-aneurysmal distal common iliac diameters between 8 and 20 mm.
10. Patient has juxtarenal aortic neck angulation ≤ 60°
11. Target branch vessel diameter ≥ 5 mm.
12. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a mycotic aneurysm or has an active systemic or local infection that may increase the risk of endovascular infection
2. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
3. Patient has a major surgical or interventional procedure, not related to the endovascular repair, planned within +/- 30 days of the AAA repair.
4. Patient has history of an aortopathic connective tissue disease (e.g. Marfan's or Ehler's-Danlos syndrome).
5. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
6. Patient has known allergy or intolerance to stainless steel, nitinol or gold (gold-coated tungsten).
7. Patient has a body habitus that would inhibit X-ray visualization of the aorta
8. Patient has a limited life expectancy of less than 1 year
9. Patient is currently participating in another investigational device or drug clinical trial
10. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
11. Thrombus or excessive calcification within the neck of the aneurysm
12. Branch vessel stenosis ≥ 80%
13. Patient treatable on label with FDA approved EVAR or FEVAR device and can wait for device availability.
14. Subject is willing and eligible to enroll in a manufacturer-sponsored study at the investigational site, or the subject is willing and eligible to participate in a study with a manufacturer-made device at another institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
All Cause Mortality | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including all-cause mortality.
Myocardial Infarction | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including myocardial infarction.
Stroke | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including stroke.
Renal Failure | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including renal failure.
Respiratory Failure | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including respiratory failure.
Paraplegia | 30 days post index procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including paraplegia.
Bowel Ischemia | 30 days post procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including bowel ischemia.
Procedural Blood Loss (>1000 cc) | 30 days post procedure
  The primary safety endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure, including procedural blood loss (>1000 cc).
Treatment Success | 12 months post index procedure
  The primary effectiveness endpoint is the proportion of subjects that achieve Treatment Success. Treatment Success is a composite endpoint assessed at 12 months that requires the following criteria to be met:
  Technical Success (at the index procedure) is defined by the following:
  1. The physician was able to insert the delivery catheter and deliver the physician modified endovascular graft to the treatment site and preserve blood flow into the vessels intended to have blood flow preserved.
  2. Freedom from Type I & III endoleaks at 12 months
  3. Freedom from stent graft migration at 12 months
  4. Freedom from aortic aneurysm enlargement at 12 months
  5. Freedom from aortic aneurysm rupture and conversion to open repair through 12 months

SECONDARY OUTCOMES:
Mortality | 30 days, 6 months, and annually through 5 years post index procedure
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including mortality.
Aneurysm related mortality | 30 days, 6 months, and annually through 5 years post index procedure
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including aneurysm related mortality.
Aneurysm Rupture | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including aneurysm rupture.
Major Adverse Events (MAE) | 30 days, 6 months, and annually through 5 years post index procedure
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including major adverse events.
Renal failure with or without permanent dialysis | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including renal failure with or without permanent dialysis.
Graft Infection | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary safety endpoints will be evaluated at 30 days, 6 months, & 12 months following the initial implant procedure and annually through 5 years, including graft infection.
Technical Success | 30 days, 6 months, and annually through 5 years post index procedure
  Secondary effectiveness endpoints will be evaluated including technical success. Technical Success (evaluated at 30-days) is a composite of the following: a. Successful access to the arterial system using remote arterial exposure, percutaneous technique, or open surgical conduits; b. Successful delivery and deployment at the intended implantation site; c. Successful side branch catheterization and placement of bridging stents with restoration and maintenance of flow in all intended target vessels; d. Successful withdrawal of the delivery system; e. Patency of all endovascular graft and stent components; f. Absence of device deformations requiring unplanned placement of an additional device; g. Absence of Type I and III endoleaks at completion angiography that extends beyond 30 days by confirmatory imaging
Stent graft migration > 10 mm | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including stent graft migration > 10 mm.
All endoleaks | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including all endoleaks.
AAA enlargement | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including AAA enlargement.
Patency related events | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including patency related events.
Device integrity failure | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be assessed including device integrity failure.
Conversion to open repair | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including conversion to open repair.
Secondary Intervention | 30 days, 6 months, and annually through 5 years post index procedure.
  Secondary effectiveness endpoints will be evaluated including secondary interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Cali Johnson, MD, EdD, Principal Investigator — University of Utah; Nathan Droz, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided